CLINICAL TRIAL: NCT00388297
Title: A Randomized Trial of Thyroxine Therapy for Subclinical Hypothyroidism or Hypothyroxinemia Diagnosed During Pregnancy
Brief Title: Thyroid Therapy for Mild Thyroid Deficiency in Pregnancy
Acronym: TSH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The George Washington University Biostatistics Center (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: HD36801-TSH; U10HD021410 (NIH); U10HD027869 (NIH); U10HD027917 (NIH); U10HD027860 (NIH); U10HD027915 (NIH); U10HD034116 (NIH); U10HD034208 (NIH); U10HD034136 (NIH); U10HD040500 (NIH); U10HD040485 (NIH); U10HD040544 (NIH); U10HD040545 (NIH); U10HD040560 (NIH); U10HD040512 (NIH); U10HD036801 (NIH); U10HD053118 (NIH)
Record Dates: First submitted 2006-10-12; First posted 2006-10-16 (Estimated); Results first posted 2019-01-30 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Subclinical Hypothyroidism; Hypothyroxinemia; Pregnancy
Keywords: Subclinical Hypothyroidism; Hypothyroxinemia; Thyroid; Pregnancy; Intellectual Development
MeSH Terms: conditions — Thyroid Diseases | interventions — Thyroxine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Levothyroxine for Subclinical Hypothyroidism (Experimental): 100 µg of Levothryoxine for participants with subclinical hypothyroidism
  Interventions: Drug: Levothyroxine
- Placebo for Levothyroxine - Subclinincal Hypothyroidism (Placebo Comparator): Placebo for Levothyroxine for participants with subclinical hypothyroidism
  Interventions: Drug: Placebo for Levothyroxine
- Levothyroxine for Hypothyroxinemia - Hypothyroxinemia (Experimental): 50 µg of Levothyroxine for participants with hypothyroxinemia
  Interventions: Drug: Levothyroxine
- Placebo for Levothyroxine (Placebo Comparator): Placebo for Levothyroxine for participants with hypothyroxinemia
  Interventions: Drug: Placebo for Levothyroxine

INTERVENTIONS:
Drug: Levothyroxine — Coded study drug is thyroxine encapsulated in a gel capsule; matching placebo contains only cellulose. Color of capsule corresponds to mcg dose level (100mcg or 25 mcg). Subjects in subclinical hypothyroidism stratum are started on 1 capsule of 100 mcg per day; subjects in hypothyroxinemia stratum are started on 2 capsules of 25 mcg per day. Thyroxine dosing adjustments for both strata are determined centrally, using an algorithm, based on results of monthly TSH or free-T4 assays. Subjects take study medication until delivery.
  Arms: Levothyroxine for Hypothyroxinemia - Hypothyroxinemia; Levothyroxine for Subclinical Hypothyroidism
Drug: Placebo for Levothyroxine
  Arms: Placebo for Levothyroxine; Placebo for Levothyroxine - Subclinincal Hypothyroidism

SUMMARY:
The purpose of this study is to determine whether treating women, who are diagnosed with a mild imbalance of thyroid hormones during pregnancy, with thyroid hormone replacement affects their children's intellectual development at 5 years of age.

DETAILED DESCRIPTION:
Published research reports have stimulated national and international controversy regarding the value of maternal thyroxine therapy given to improve neurodevelopment of the fetus in women with variously defined hypothyroidism. These reports have led to conflicting and confusing recommendations as to whether or not all pregnant women in the U.S. should be screened for subclinical hypothyroidism or hypothyroxinemia.

Pregnant women less than 20 weeks gestation will have a blood test to screen for subclinical hypothyroidism or hypothyroxinemia. If eligible for the trial, patients will receive levothyroxine or placebo until delivery. Blood draws will be done at monthly study visits and the dosage will be adjusted based on test results. The children of these patients will have developmental testing done annually until they are 5 years of age.

Comparison(s): thyroxine supplementation versus placebo given during pregnancy to determine whether therapy is effective in improving intellectual ability at 5 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Subclinical Hypothyroidism as defined by an elevated TSH (≥ 3.00 mU/L) and a free-T4 in the normal range (i.e. 0.86 to 1.90 ng/dL) or Hypothyroxinemia as defined by a TSH in the normal range (0.08 to 2.99 micrometers (mU)/L) and a low free-T4 (<0.86 ng/dL)
* Singleton Pregnancy
* Gestational age at randomization between 8 weeks 0 days and 20 weeks 6 days

Exclusion Criteria:

1. Major fetal anomaly or demise
2. Planned termination of the pregnancy
3. History of thyroid cancer or current thyroid disease requiring medication
4. Diabetes, on medication (insulin, glyburide)
5. Collagen vascular disease (autoimmune disease), such as lupus, scleroderma and polymyalgia rheumatica, on medication
6. Receiving anticoagulant therapy
7. Depression, currently on treatment with tricyclics or selective serotonin reuptake inhibitors (SSRIs)
8. Other known serious maternal medical complications including:

   1. Chronic hypertension requiring antihypertensive medication (including diuretics)
   2. Epilepsy or other seizure disorder, on medication
   3. Active or chronic liver disease (acute hepatitis, chronic active hepatitis) with persistently abnormal liver enzymes
   4. Cancer (including melanoma but excluding other skin cancers)
   5. Heart disease (tachyrhythmia, class II or greater heart disease or on heart medication). Mitral valve prolapse without arrhythmia is not an exclusion.
   6. Asthma, on oral corticosteroids
9. Known illicit drug or alcohol abuse during current pregnancy
10. Delivery at a non-network hospital
11. Participation in another intervention study that influences maternal and fetal morbidity and mortality, or participation in this trial in a previous pregnancy
12. Unwilling or unable to commit to 5 year follow-up of the infant

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1203 (Actual)
Dates: Start 2006-10; Primary Completion 2015-08 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Casey, MD, Study Chair — University of Texas Southwestern Medical Center; Menachem Miodovnik, MD, Study Director — NICHD Project Scientist
Locations (14):
- United States (14):
  - University of Alabama - Birmingham, Birmingham, Alabama
  - Northwestern University, Chicago, Illinois
  - Wayne State University, Detroit, Michigan
  - Columbia University, New York, New York
  - University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Case Western University, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Oregon Health & Sciences University, Portland, Oregon
  - University of Pittsburgh Magee Womens Hospital, Pittsburgh, Pennsylvania
  - Brown University, Providence, Rhode Island
  - University of Texas - Southwest, Dallas, Texas
  - University of Texas Medical Branch - Galveston, Galveston, Texas
  - University of Texas-Houston, Houston, Texas
  - University of Utah Medical Center, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
The data will be shared after the completion of the trial and publication of the main analyses per NIH policy. When made available, requests for the dataset(s) can be sent to mfmudatasets@bsc.gwu.edu.

REFERENCES:
- [Derived] Smid MC, Metz TD, McMillin GA, Mele L, Casey BM, Reddy UM, Wapner RJ, Thorp JM, Saade GR, Tita ATN, Miller ES, Rouse DJ, Sibai B, Costantine MM, Mercer BM, Caritis SN; for the Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) Maternal-Fetal Medicine Units (MFMU) Network*. Prenatal Nicotine or Cannabis Exposure and Offspring Neurobehavioral Outcomes. Obstet Gynecol. 2022 Jan 1;139(1):21-30. doi: 10.1097/AOG.0000000000004632. PMID 34856574
- [Derived] Casey BM, Thom EA, Peaceman AM, Varner MW, Sorokin Y, Hirtz DG, Reddy UM, Wapner RJ, Thorp JM Jr, Saade G, Tita AT, Rouse DJ, Sibai B, Iams JD, Mercer BM, Tolosa J, Caritis SN, VanDorsten JP; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Treatment of Subclinical Hypothyroidism or Hypothyroxinemia in Pregnancy. N Engl J Med. 2017 Mar 2;376(9):815-825. doi: 10.1056/NEJMoa1606205. PMID 28249134
- See also: Click here for more information about this study — http://www.bsc.gwu.edu/mfmu/Projects/Projects.cgi

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled women with a singleton pregnancy before 20 weeks gestation who met the criteria for either subclinical hypothyroidism or hypothyroxinemia based on serum thyrotropin and free T4 values. The study was conducted as two multicenter, randomized, placebo-controlled trials at 15 NICHD MFMU network centers.
Pre-assignment Details: 97,228 patients were screened during the recruitment period October 2006 to October 2009, Of the 800 eligible based on subclinical hypothyroidism, 677 completed the 7-day placebo adherence run-in and were randomized. Of the 632 eligible based on hypothyroxinemia, 526 completed the run-in phase and were randomized.
Groups:
- Levothyroxine for Subclinical Hypothyroidism; Levothyroxine for Hypothyroxinemia: Levothyroxine
  Levothyroxine: Coded study drug is thyroxine encapsulated in a gel capsule; matching placebo contains only cellulose. Color of capsule corresponds to mcg dose level (100mcg or 25 mcg). Subjects in subclinical hypothyroidism stratum are started on 1 capsule of 100 mcg per day; subjects in hypothyroxinemia stratum are started on 2 capsules of 25 mcg per day. Thyroxine dosing adjustments for both strata are determined centrally, using an algorithm, based on results of monthly TSH or free-T4 assays. Subjects take study medication until delivery.
- Placebo for Levothyroxine - Subclinical Hypothyroidism: Placebo for Levothyroxine for the Subclinical Hypothyroidism group
- Placebo for Levothyroxine for Hypothyroxinemia: Placebo for Levothyroxine for the Hypothyroxinemia group
Period: Overall Study
Arm/Group | Levothyroxine for Subclinical Hypothyroidism | Placebo for Levothyroxine - Subclinical Hypothyroidism | Levothyroxine for Hypothyroxinemia | Placebo for Levothyroxine for Hypothyroxinemia
Started | 339 | 338 | 265 | 261
Completed | 323 | 326 | 254 | 253
Not Completed | 16 | 12 | 11 | 8
Not completed — Lost to Follow-up | 16 | 12 | 11 | 8

BASELINE CHARACTERISTICS:
Groups:
- Placebo for Levothyroxine - Subclinical Hypothyroidism: Placebo for Levothyroxine for the Subclinical Hypothyroidism
- Placebo for Levothyroxine - Hypothyroxinemia: Placebo for Levothyroxine for the Hypothyroxinemia
- Total: Total of all reporting groups
Arm/Group | Levothyroxine for Subclinical Hypothyroidism | Placebo for Levothyroxine - Subclinical Hypothyroidism | Levothyroxine for Hypothyroxinemia | Placebo for Levothyroxine - Hypothyroxinemia | Total
Number analyzed (Participants) | 339 | 338 | 265 | 261 | 1203
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.7 (5.7) | 27.3 (5.7) | 27.8 (5.7) | 28.0 (5.8) | 27.7 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 339 | 338 | 265 | 261 | 1203
  Male | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 27 | 25 | 61 | 65 | 178
  Hispanic | 195 | 185 | 131 | 125 | 636
  White | 109 | 117 | 69 | 69 | 364
  Other | 8 | 11 | 4 | 2 | 25
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 339 | 338 | 265 | 261 | 1203
Body-mass index [Mean (Standard Deviation); unit: kg/m^2] | 28.1 (6.4) | 28.2 (6.4) | 30.3 (6.4) | 30.2 (7.1) | 29.0 (6.6)
Nulliparous [Count of Participants; unit: Participants] | 124 | 134 | 69 | 64 | 391
Baseline thyrotropin (mU/liter) Median [Median (Inter-Quartile Range); unit: mU/liter] | 4.5 [4.0 to 5.5] | 4.3 [4.0 to 5.3] | 1.5 [1.1 to 2.1] | 1.4 [1.0 to 2.1] | 3.4 [1.6 to 4.6]
Baseline free thyroxine (ng/dl Median [Median (Inter-Quartile Range); unit: ng/dl] | 1.01 [.94 to 1.09] | 1.02 [0.96 to 1.11] | 0.83 [0.81 to 0.84] | 0.83 [0.81 to 0.84] | 0.90 [0.83 to 1.03]
Urinary iodine (µg/liter) Median [Median (Inter-Quartile Range); unit: µg/liter] | 199 [106 to 340] | 196 [114 to 331] | 185 [108 to 341] | 191 [118 to 325] | 194 [111 to 334]
Weeks Gestation at Randomization [Mean (Standard Deviation); unit: Weeks] | 16.6 (3.0) | 16.7 (3.0) | 18.0 (2.8) | 17.7 (2.9) | 17.2 (3.0)

OUTCOME MEASURES:

1. Primary Outcome: Intellectual Function of Children at 5 Years of Age in Women Diagnosed With a) Subclinical Hypothyroidism or b) Hypothyroxinemia During the First Half of Pregnancy, or Death.
Description: The primary outcome was death or IQ score at 5 years of age (or at 3 years of age if the 5-year examination was missing). The full-scale IQ was assessed with the use of the Wechsler Preschool and Primary Scale of Intelligence III (WPPSI-III) at 5 years of age or the overall (general conceptual ability) score from the Differential Ability Scales-II at 3 years of age if the WPPSI-III score was not available. Results are expressed as an age-standardized score, with an expected population mean of 100 and a standard deviation of 15. Death before 3 years of age was assigned a score of 0 (lowest possible rank) and was included in the estimation of the median.
  For Quotient and Composite score:
  below 70 is Extremely Low, 70-79 is Borderline, 80-89 is Low Average, 90-109 is Average, 110-119 is High Average, 120-129 is Superior, 130+
Time Frame: 60 months of age
Measure: Median (95% Confidence Interval); unit: score on a scale
Arm/Group | Levothyroxine for Subclinical Hypothyroidism | Placebo for Levothyroxine - Subclinical Hypothyroidism | Levothyroxine for Hypothyroxinemia | Placebo for Levothyroxine - Hypothyroxinemia
Number analyzed (Participants) | 323 | 326 | 254 | 253
score on a scale | 97 [94 to 99] | 94 [92 to 96] | 94 [91 to 95] | 91 [89 to 93]
Statistical Analysis 1: Comparison: Levothyroxine for Subclinical Hypothyroidism vs Placebo for Levothyroxine - Subclinical Hypothyroidism; Test type: Superiority or Other; p = 0.71, Wilcoxon (Mann-Whitney); Hodges-Lehmann estimate = 0, 95% CI 2-sided [-3 to 2]
Statistical Analysis 2: Comparison: Levothyroxine for Hypothyroxinemia vs Placebo for Levothyroxine - Hypothyroxinemia; Test type: Superiority or Other; p = 0.30, Wilcoxon (Mann-Whitney); Hodges-Lehmann estimate = -1, 95% CI 2-sided [-4 to 1]

2. Secondary Outcome: Week of Gestation at Delivery
Description: Gestational age at delivery and preterm birth < 37 weeks' gestation or < 34 weeks' gestation
Time Frame: Delivery
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Levothyroxine for Subclinical Hypothyroidism | Placebo for Levothyroxine - Subclinical Hypothyroidism | Levothyroxine for Hypothyroxinemia | Placebo for Levothyroxine - Hypothyroxinemia
Number analyzed (Participants) | 339 | 338 | 263 | 261
weeks | 39.1 (2.5) | 38.9 (3.1) | 39.0 (2.4) | 38.8 (3.1)
Statistical Analysis 1: Comparison: Levothyroxine for Subclinical Hypothyroidism vs Placebo for Levothyroxine - Subclinical Hypothyroidism; Test type: Superiority or Other; p = 0.57, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Levothyroxine for Hypothyroxinemia vs Placebo for Levothyroxine - Hypothyroxinemia; Test type: Superiority or Other; p = 0.46, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Number of Participants With Preterm Delivery
Description: Preterm delivery at less than 37 weeks or less than 34 weeks gestation
Time Frame: Delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Levothyroxine for Subclinical Hypothyroidism | Placebo for Levothyroxine - Subclinical Hypothyroidism | Levothyroxine for Hypothyroxinemia | Placebo for Levothyroxine - Hypothyroxinemia
Number analyzed (Participants) | 339 | 338 | 263 | 261
Participants
  Preterm birth < 34 wk | 9 | 10 | 10 | 7
  Preterm birth < 37 wk | 31 | 37 | 31 | 20
Statistical Analysis 1: Comparison: Levothyroxine for Subclinical Hypothyroidism vs Placebo for Levothyroxine - Subclinical Hypothyroidism; Analysis for < 34 weeks; Test type: Superiority or Other; p = 0.81, Chi-squared
Statistical Analysis 2: Comparison: Levothyroxine for Hypothyroxinemia vs Placebo for Levothyroxine - Hypothyroxinemia; Analysis for <34 weeks; Test type: Superiority or Other; p = 0.47, Chi-squared
Statistical Analysis 3: Comparison: Levothyroxine for Subclinical Hypothyroidism vs Placebo for Levothyroxine - Subclinical Hypothyroidism; Analysis for <37 weeks; Test type: Superiority or Other; p = 0.44, Chi-squared
Statistical Analysis 4: Comparison: Levothyroxine for Hypothyroxinemia vs Placebo for Levothyroxine - Hypothyroxinemia; Analysis for < 37 weeks; Test type: Superiority or Other; p = 0.11, Chi-squared
Statistical Analysis 5: Comparison: Levothyroxine for Subclinical Hypothyroidism vs Placebo for Levothyroxine - Subclinical Hypothyroidism; Bayley-III Motor (24 months); Test type: Superiority or Other; p = 0.31, Chi-squared; Hodges-Lehmann = 0, 95% CI 2-sided [0 to 3]
Statistical Analysis 6: Comparison: Levothyroxine for Subclinical Hypothyroidism vs Placebo for Levothyroxine - Subclinical Hypothyroidism; Bayley-II Language (24 months); Test type: Superiority or Other; p = 0.30, Chi-squared; Hodges-Lehmann = 0, 95% CI 2-sided [0 to 3]
Statistical Analysis 7: Comparison: Levothyroxine for Hypothyroxinemia vs Placebo for Levothyroxine - Hypothyroxinemia; Bayley-III Cognitive (12 months); Test type: Superiority or Other; p = 0.89, Chi-squared; Hodges-Lehmann = 0, 95% CI 2-sided [0 to 0]
Statistical Analysis 8: Comparison: Levothyroxine for Hypothyroxinemia vs Placebo for Levothyroxine - Hypothyroxinemia; Bayley-III Motor (12 months); Test type: Superiority or Other; p = 0.54, Chi-squared; Hodges-Lehmann = 0, 95% CI 2-sided [0 to 3]
Statistical Analysis 9: Comparison: Levothyroxine for Hypothyroxinemia vs Placebo for Levothyroxine - Hypothyroxinemia; Bayley-III Language (12 months); Test type: Superiority or Other; p = 0.92, Chi-squared; Hodges-Lehmann = 0, 95% CI 2-sided [-3 to 3]
Statistical Analysis 10: Comparison: Levothyroxine for Hypothyroxinemia vs Placebo for Levothyroxine - Hypothyroxinemia; Bayley-III Cognitive (24 months); Test type: Superiority or Other; p = 0.70, Chi-squared; Hodges-Lehmann = 0, 95% CI 2-sided [0 to 0]
Statistical Analysis 11: Comparison: Levothyroxine for Hypothyroxinemia vs Placebo for Levothyroxine - Hypothyroxinemia; Bayley-III Motor (24 months); Test type: Superiority or Other; p = 0.20, Chi-squared; Hodges-Lehmann = 0, 95% CI 2-sided [-3 to 0]
Statistical Analysis 12: Comparison: Levothyroxine for Hypothyroxinemia vs Placebo for Levothyroxine - Hypothyroxinemia; Bayley-II Language (24 months); Test type: Superiority or Other; p = 0.71, Chi-squared; Hodges-Lehmann = 0, 95% CI 2-sided [-3 to 2]

4. Secondary Outcome: Selected Cognitive Abilities From the Subscales of the Wechsler Preschool and Primary Scale of Intelligence (WPPSI-III)
Description: Standardized full-scale IQ scores from the Wechsler Preschool and Primary Scale of Intelligence III (WPPSI-III) at 5 years of age. Quotient and Composite scores have a mean of 100 and a standard deviation of 15. Subtest scaled scores have a mean of 10 and a standard deviation of 3.
  For Quotient and Composite score:
  below 70 is Extremely Low, 70-79 is Borderline, 80-89 is Low Average, 90-109 is Average, 110-119 is High Average, 120-129 is Superior, 130+ is Very Superior.
Time Frame: 60 months
Measure: Median (95% Confidence Interval); unit: score on a scale
Arm/Group | Levothyroxine for Subclinical Hypothyroidism | Placebo for Levothyroxine - Subclinical Hypothyroidism | Levothyroxine for Hypothyroxinemia | Placebo for Levothyroxine - Hypothyroxinemia
Number analyzed (Participants) | 311 | 314 | 243 | 243
score on a scale | 97 [95 to 99] | 95 [93 to 97] | 94 [91 to 95] | 92 [90 to 95]
Statistical Analysis 1: Comparison: Levothyroxine for Subclinical Hypothyroidism vs Placebo for Levothyroxine - Subclinical Hypothyroidism; Test type: Superiority or Other; p = 0.89, Chi-squared; Hodges-Lehmann = 0, 95% CI 2-sided [-3 to 2]
Statistical Analysis 2: Comparison: Levothyroxine for Hypothyroxinemia vs Placebo for Levothyroxine - Hypothyroxinemia; Test type: Superiority or Other; p = 0.48, Chi-squared; Hodges-Lehmann = -1, 95% CI 2-sided [-3 to 2]

5. Secondary Outcome: Cognitive and Achievement Levels From the Differential Ability Scales (DAS II)
Description: Overall general conceptual ability score as measured by the DAS-II at 36 months of age.
  GCA General Conceptual Ability Classification ≥ 130 Very high 120-129 High 110-119 Above average 90-109 Average 80-89 Below average 70-79 Low
  ≤ 69 Very low
Time Frame: 36 months
Measure: Median (95% Confidence Interval); unit: score on a scale
Arm/Group | Levothyroxine for Subclinical Hypothyroidism | Placebo for Levothyroxine - Subclinical Hypothyroidism | Levothyroxine for Hypothyroxinemia | Placebo for Levothyroxine - Hypothyroxinemia
Number analyzed (Participants) | 304 | 308 | 244 | 235
score on a scale | 90 [88 to 93] | 90 [87 to 93] | 90 [87 to 92] | 89 [87 to 91]
Statistical Analysis 1: Comparison: Levothyroxine for Subclinical Hypothyroidism vs Placebo for Levothyroxine - Subclinical Hypothyroidism; Test type: Superiority or Other; p = 0.90, Chi-squared; Hodges-Lehmann = 0, 95% CI 2-sided [-2 to 3]
Statistical Analysis 2: Comparison: Levothyroxine for Hypothyroxinemia vs Placebo for Levothyroxine - Hypothyroxinemia; Test type: Superiority or Other; p = 0.64, Chi-squared; Hodges-Lehmann = -1, 95% CI 2-sided [-3 to 2]

6. Secondary Outcome: Cognitive and Achievement Levels From Two DAS-II Subtests (Recall of Digits Forward and Recognition of Pictures)
Description: Cognitive and achievement levels from two DAS-II subtests (Recall of Digits Forward and Recognition of Pictures)
  GCA General Conceptual Ability Classification ≥ 130 Very high 120-129 High 110-119 Above average 90-109 Average 80-89 Below average 70-79 Low
  ≤ 69 Very low
Time Frame: 48 months of age
Population: For all outcomes except the primary outcome, the potential follow-up cohort consisted of 335 children in the levothyroxine group and 329 in the placebo group for the mothers with subclinical hypothyroidism and for the hypothyroxinemia group - 260 children in the levothyroxine group and 255 children in the placebo group.
Measure: Median (95% Confidence Interval); unit: score on a scale
Arm/Group | Levothyroxine for Subclinical Hypothyroidism | Placebo for Levothyroxine - Subclinical Hypothyroidism | Levothyroxine for Hypothyroxinemia | Placebo for Levothyroxine - Hypothyroxinemia
Number analyzed (Participants) | 335 | 329 | 260 | 255
score on a scale
  Median Recall of Digits Forward Score: number analyzed (Participants) | 298 | 299 | 236 | 224
  Median Recall of Digits Forward Score | 84 [76 to 91] | 84 [76 to 91] | 91 [84 to 99] | 74 [74 to 80]
  Median Recognition of Pictures Score: number analyzed (Participants) | 298 | 302 | 234 | 226
  Median Recognition of Pictures Score | 74 [74 to 80] | 74 [74 to 80] | 84 [84 to 91] | 74 [74 to 80]
Statistical Analysis 1: Comparison: Levothyroxine for Subclinical Hypothyroidism vs Placebo for Levothyroxine - Subclinical Hypothyroidism; Analysis for recall of digits forward; Test type: Superiority or Other; p = 0.60, Chi-squared; Hodges-Lehmann = 0, 95% CI 2-sided [-5 to 7]
Statistical Analysis 2: Comparison: Levothyroxine for Hypothyroxinemia vs Placebo for Levothyroxine - Hypothyroxinemia; Analysis for recall of digits forward; Test type: Superiority or Other; p = 0.22, Chi-squared; Hodges-Lehmann = 0, 95% CI 2-sided [-8 to 0]
Statistical Analysis 3: Comparison: Levothyroxine for Subclinical Hypothyroidism vs Placebo for Levothyroxine - Subclinical Hypothyroidism; Analysis for Recognition of Pictures; Test type: Superiority or Other; p = 0.52, Chi-squared; Hodges-Lehmann = 0, 95% CI 2-sided [-6 to 0]
Statistical Analysis 4: Comparison: Levothyroxine for Hypothyroxinemia vs Placebo for Levothyroxine - Hypothyroxinemia; Analysis for Recognition of Pictures; Test type: Superiority or Other; p = 0.91, Chi-squared; Hodges-Lehmann = 0, 95% CI 2-sided [-4 to 0]

7. Secondary Outcome: Cognitive, Motor and Language Scale Scores From the Bayley Certified Scales of Infant Development III Edition
Description: Composite scores are derived for cognitive, language, and motor development and scaled to a metric, with a mean of 100, standard deviation of 15, and range of 40 to 160. Results can also be expressed as percentile ranks relative to the standardization sample, with a mean and median of 50 and range from 1 to 99
Time Frame: 12 and 24 months of age
Population: For all outcomes except the primary outcome the potential follow-up cohort in the subclinical hypothyroidism groups consisted of 335 children in the levothyroxine group and 329 in the placebo group, and for the hypothyroxinema groups: 254 children in the levothryoxine group and 253 children in the placebo group.
Measure: Median (95% Confidence Interval); unit: score on a scale
Arm/Group | Levothyroxine for Subclinical Hypothyroidism | Placebo for Levothyroxine - Subclinical Hypothyroidism | Levothyroxine for Hypothyroxinemia | Placebo for Levothyroxine - Hypothyroxinemia
Number analyzed (Participants) | 323 | 326 | 254 | 253
score on a scale
  Median 12 mo cognitive score: number analyzed (Participants) | 311 | 315 | 247 | 238
  Median 12 mo cognitive score | 100 [95 to 100] | 100 [95 to 100] | 100 [100 to 100] | 100 [100 to 100]
  Median 12 mo motor score: number analyzed (Participants) | 312 | 314 | 246 | 236
  Median 12 mo motor score | 97 [97 to 97] | 97 [97 to 97] | 97 [94 to 97] | 97 [94 to 97]
  Median 12 mo language score: number analyzed (Participants) | 309 | 312 | 246 | 237
  Median 12 mo language score | 94 [94 to 97] | 94 [94 to 97] | 94 [91 to 94] | 94 [91 to 94]
  Median 24 mo cognitive score: number analyzed (Participants) | 308 | 302 | 235 | 235
  Median 24 mo cognitive score | 90 [90 to 90] | 90 [90 to 90] | 90 [85 to 90] | 90 [85 to 90]
  Median 24 mo motor score: number analyzed (Participants) | 304 | 300 | 233 | 232
  Median 24 mo motor score | 97 [97 to 97] | 97 [97 to 100] | 97 [94 to 100] | 97 [94 to 97]
  Median 24 mo language score: number analyzed (Participants) | 300 | 296 | 232 | 229
  Median 24 mo language score | 89 [89 to 91] | 91 [89 to 94] | 89 [89 to 94] | 89 [89 to 94]
Statistical Analysis 1: Comparison: Levothyroxine for Subclinical Hypothyroidism vs Placebo for Levothyroxine - Subclinical Hypothyroidism; Bayley II Cognitive (12 months); Test type: Superiority or Other; p = 0.63, Chi-squared; Hodges-Lehmann = 0, 95% CI 2-sided [0 to 0]
Statistical Analysis 2: Comparison: Levothyroxine for Subclinical Hypothyroidism vs Placebo for Levothyroxine - Subclinical Hypothyroidism; Bayley II Motor (12 mo); Test type: Superiority or Other; p = 0.83, Chi-squared; Hodges-Lehmann = 0, 95% CI 2-sided [0 to 3]
Statistical Analysis 3: Comparison: Levothyroxine for Subclinical Hypothyroidism vs Placebo for Levothyroxine - Subclinical Hypothyroidism; Bayley-III Language (12 months); Test type: Superiority or Other; p = 0.48, Chi-squared; Hodges-Lehmann = 0, 95% CI 2-sided [0 to 3]
Statistical Analysis 4: Comparison: Levothyroxine for Subclinical Hypothyroidism vs Placebo for Levothyroxine - Subclinical Hypothyroidism; Bayley-III Cognitive (24 months); Test type: Superiority or Other; p = 0.59, Chi-squared; Hodges-Lehmann = 0, 95% CI 2-sided [0 to 0]

8. Secondary Outcome: Behavioral Problems and Social Competencies at 36 and 60 Months of Age, as Measured by the Child Behavior Checklist (CBCL)
Description: Behavioral problems and social competencies at 36 and 60 months of age, as measured by the Child Behavior Checklist (CBCL). The CBCL is filled out by the caregiver. Each of the 100 questions indicates a behavior for which the caregiver scores as Not True (0), Sometimes True (1), or Often True (2). The scores for all the questions are then summed and evaluated against the normative data/T-scores. A Tscore of less than 60 is considered to be in the normal range. A T score of 60-63 is a borderline, and a T score of more than 63 is in the clinical range. Lower scores represent better outcomes.
Time Frame: 36 and 60 months of age
Population: The potential follow-up cohort consisted of 335 children in the levothyroxine group and 329 in the placebo group for subclinical hypothyroidism and for hypothyroxinemia - 260 children in the levothyroxine group and 255 in the placebo group. A Child Behavior Checklist T score of less than 60 is considered to be in the normal range.
Measure: Median (95% Confidence Interval); unit: T-score
Arm/Group | Levothyroxine for Subclinical Hypothyroidism | Placebo for Levothyroxine - Subclinical Hypothyroidism | Levothyroxine for Hypothyroxinemia | Placebo for Levothyroxine - Hypothyroxinemia
Number analyzed (Participants) | 335 | 314 | 260 | 255
T-score
  CBCL T score at 36 mo: number analyzed (Participants) | 306 | 309 | 244 | 237
  CBCL T score at 36 mo | 46 [45 to 48] | 46 [45 to 48] | 48 [46 to 50] | 48 [45 to 49]
  CBCL T score at 60 mo: number analyzed (Participants) | 314 | 313 | 244 | 243
  CBCL T score at 60 mo | 44 [43 to 46] | 44 [42 to 46] | 45 [43 to 46] | 43 [42 to 45]
Statistical Analysis 1: Comparison: Levothyroxine for Subclinical Hypothyroidism vs Placebo for Levothyroxine - Subclinical Hypothyroidism; CBCL at 36 months; Test type: Superiority or Other; p = 0.99, Chi-squared; Hodges-Lehmann = 0, 95% CI 2-sided [-2 to 2]
Statistical Analysis 2: Comparison: Levothyroxine for Subclinical Hypothyroidism vs Placebo for Levothyroxine - Subclinical Hypothyroidism; CBCL at 60 months; Test type: Superiority or Other; p = 0.96, Chi-squared; Hodges-Lehmann = 0, 95% CI 2-sided [-2 to 2]
Statistical Analysis 3: Comparison: Levothyroxine for Hypothyroxinemia vs Placebo for Levothyroxine - Hypothyroxinemia; CBCL at 36 months; Test type: Superiority or Other; p = 0.65, Chi-squared; Hodges-Lehmann = 0, 95% CI 2-sided [-2 to 2]
Statistical Analysis 4: Comparison: Levothyroxine for Hypothyroxinemia vs Placebo for Levothyroxine - Hypothyroxinemia; CBCL at 60 months; Test type: Superiority or Other; p = 0.44, Chi-squared; Hodges-Lehmann = -1, 95% CI 2-sided [-3 to 1]

9. Secondary Outcome: Attention Deficit Hyperactivity Disorder (ADHD) Index Score From the Connors' Rating Scales (Parent-S) - Revised
Description: The Conners' Rating Scales-Revised were used to assess attention deficit-hyperactivity disorder (ADHD). A T score of 45 to 55 is considered to be typical or average; a T score of 44 or less is not a concern, a T score of 56 to 60 is considered to be a borderline score, and a T score of 61 or higher indicates a possible or clinically significant problem.
Time Frame: 48 months of age
Measure: Median (95% Confidence Interval); unit: T-score
Arm/Group | Levothyroxine for Subclinical Hypothyroidism | Placebo for Levothyroxine - Subclinical Hypothyroidism | Levothyroxine for Hypothyroxinemia | Placebo for Levothyroxine - Hypothyroxinemia
Number analyzed (Participants) | 302 | 303 | 238 | 228
T-score | 48 [47 to 49] | 49 [47 to 51] | 50 [49 to 51] | 49 [48 to 51]
Statistical Analysis 1: Comparison: Levothyroxine for Subclinical Hypothyroidism vs Placebo for Levothyroxine - Subclinical Hypothyroidism; Test type: Superiority or Other; p = 0.37, Chi-squared; Hodges-Lehmann = 0, 95% CI 2-sided [-1 to 2]
Statistical Analysis 2: Comparison: Levothyroxine for Hypothyroxinemia vs Placebo for Levothyroxine - Hypothyroxinemia; Test type: Superiority or Other; p = 0.98, Chi-squared; Hodges-Lehmann = 0, 95% CI 2-sided [-2 to 2]

10. Secondary Outcome: Participants With Placental Abruption
Description: Clinically significant placental abruption will be determined by centralized (blinded) chart review
Time Frame: Duration of pregnancy, delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Levothyroxine for Subclinical Hypothyroidism | Placebo for Levothyroxine - Subclinical Hypothyroidism | Levothyroxine for Hypothyroxinemia | Placebo for Levothyroxine - Hypothyroxinemia
Number analyzed (Participants) | 339 | 338 | 263 | 261
Participants | 1 | 5 | 3 | 2
Statistical Analysis 1: Comparison: Levothyroxine for Subclinical Hypothyroidism vs Placebo for Levothyroxine - Subclinical Hypothyroidism; Test type: Superiority or Other; p = 0.12, Chi-squared
Statistical Analysis 2: Comparison: Levothyroxine for Hypothyroxinemia vs Placebo for Levothyroxine - Hypothyroxinemia; Test type: Superiority or Other; p = 1.00, Chi-squared

11. Secondary Outcome: Participants With Gestational Hypertension
Description: Gestational hypertension defined as patient having a diastolic ≥ 90 during pregnancy without proteinuria
Time Frame: During pregnancy and until delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Levothyroxine for Subclinical Hypothyroidism | Placebo for Levothyroxine - Subclinical Hypothyroidism | Levothyroxine for Hypothyroxinemia | Placebo for Levothyroxine - Hypothyroxinemia
Number analyzed (Participants) | 339 | 338 | 263 | 261
Participants | 33 | 36 | 20 | 24
Statistical Analysis 1: Comparison: Levothyroxine for Subclinical Hypothyroidism vs Placebo for Levothyroxine - Subclinical Hypothyroidism; Test type: Superiority or Other; p = 0.69, Chi-squared
Statistical Analysis 2: Comparison: Levothyroxine for Hypothyroxinemia vs Placebo for Levothyroxine - Hypothyroxinemia; Test type: Superiority or Other; p = 0.51, Chi-squared

12. Secondary Outcome: Participants With Preeclampsia
Description: Preeclampsia defined as patient having a diastolic ≥ 90 during pregnancy with at least 1 + proteinuria. Preeclampsia will also include HELLP syndrome or eclampsia.
Time Frame: Duration of pregnancy, Delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Levothyroxine for Subclinical Hypothyroidism | Placebo for Levothyroxine - Subclinical Hypothyroidism | Levothyroxine for Hypothyroxinemia | Placebo for Levothyroxine - Hypothyroxinemia
Number analyzed (Participants) | 339 | 338 | 263 | 261
Participants | 22 | 20 | 9 | 11
Statistical Analysis 1: Comparison: Levothyroxine for Subclinical Hypothyroidism vs Placebo for Levothyroxine - Subclinical Hypothyroidism; Test type: Superiority or Other; p = 0.76, Chi-squared
Statistical Analysis 2: Comparison: Levothyroxine for Hypothyroxinemia vs Placebo for Levothyroxine - Hypothyroxinemia; Test type: Superiority or Other; p = 0.64, Chi-squared

13. Secondary Outcome: Gestational Diabetes Mellitus
Description: A patient is considered to have gestational diabetes if clinically diagnosed with class A1 or A2
Time Frame: During pregnancy until delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Levothyroxine for Subclinical Hypothyroidism | Placebo for Levothyroxine - Subclinical Hypothyroidism | Levothyroxine for Hypothyroxinemia | Placebo for Levothyroxine - Hypothyroxinemia
Number analyzed (Participants) | 339 | 338 | 263 | 261
Participants | 25 | 22 | 21 | 24
Statistical Analysis 1: Comparison: Levothyroxine for Subclinical Hypothyroidism vs Placebo for Levothyroxine - Subclinical Hypothyroidism; Test type: Superiority or Other; p = 0.66, Chi-squared
Statistical Analysis 2: Comparison: Levothyroxine for Hypothyroxinemia vs Placebo for Levothyroxine - Hypothyroxinemia; Test type: Superiority or Other; p = 0.62, Chi-squared

14. Secondary Outcome: Participants With Composite Neonatal Outcome
Description: The composite neonatal outcome was defined as periventricular leukomalacia, intraventricular hemorrhage of grade III or IV, necrotizing enterocolitis (stage ≥II), severe retinopathy of prematurity (stage ≥III), the severe respiratory distress syndrome, bronchopulmonary dysplasia, neonatal death, stillbirth, or serious infectious complication.
Time Frame: Within 72 hours of delivery.
Measure: Count of Participants; unit: Participants
Arm/Group | Levothyroxine for Subclinical Hypothyroidism | Placebo for Levothyroxine - Subclinical Hypothyroidism | Levothyroxine for Hypothyroxinemia | Placebo for Levothyroxine - Hypothyroxinemia
Number analyzed (Participants) | 339 | 338 | 263 | 261
Participants | 7 | 12 | 5 | 7
Statistical Analysis 1: Comparison: Levothyroxine for Subclinical Hypothyroidism vs Placebo for Levothyroxine - Subclinical Hypothyroidism; Test type: Superiority or Other; p = 0.24, Chi-squared
Statistical Analysis 2: Comparison: Levothyroxine for Hypothyroxinemia vs Placebo for Levothyroxine - Hypothyroxinemia; Test type: Superiority or Other; p = 0.55, Chi-squared

15. Secondary Outcome: Participants Who Experienced a Stillbirth or Miscarriage
Description: Stillbirth or miscarriage.
Time Frame: Delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Levothyroxine for Subclinical Hypothyroidism | Placebo for Levothyroxine - Subclinical Hypothyroidism | Levothyroxine for Hypothyroxinemia | Placebo for Levothyroxine - Hypothyroxinemia
Number analyzed (Participants) | 339 | 338 | 263 | 261
Participants | 4 | 7 | 2 | 5
Statistical Analysis 1: Comparison: Levothyroxine for Subclinical Hypothyroidism vs Placebo for Levothyroxine - Subclinical Hypothyroidism; Test type: Superiority or Other; p = 0.36, Chi-squared
Statistical Analysis 2: Comparison: Levothyroxine for Hypothyroxinemia vs Placebo for Levothyroxine - Hypothyroxinemia; Test type: Superiority or Other; p = 0.28, Chi-squared

16. Secondary Outcome: Number of Neonatal Deaths
Description: Fetal and neonatal death
Time Frame: Through 72 hours post delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Levothyroxine for Subclinical Hypothyroidism | Placebo for Levothyroxine - Subclinical Hypothyroidism | Levothyroxine for Hypothyroxinemia | Placebo for Levothyroxine - Hypothyroxinemia
Number analyzed (Participants) | 339 | 338 | 263 | 261
Participants | 0 | 1 | 1 | 1
Statistical Analysis 1: Comparison: Levothyroxine for Subclinical Hypothyroidism vs Placebo for Levothyroxine - Subclinical Hypothyroidism; Test type: Superiority or Other; p = 0.50, Chi-squared
Statistical Analysis 2: Comparison: Levothyroxine for Hypothyroxinemia vs Placebo for Levothyroxine - Hypothyroxinemia; Test type: Superiority or Other; p = 1.00, Chi-squared

17. Secondary Outcome: Number of Infants With Apgar Score 4 at 1 Minute and < 7 at 5 Minutes
Description: Apgar score < 4 at 1 minute and < 7 at 5 minutes
Time Frame: 1 minute and 5 minutes post delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Levothyroxine for Subclinical Hypothyroidism | Placebo for Levothyroxine - Subclinical Hypothyroidism | Levothyroxine for Hypothyroxinemia | Placebo for Levothyroxine - Hypothyroxinemia
Number analyzed (Participants) | 339 | 338 | 263 | 261
Participants
  Apgar < 4 at 1 minute | 6 | 7 | 6 | 7
  Apgar < 7 at 5 minutes | 2 | 3 | 2 | 4
Statistical Analysis 1: Comparison: Levothyroxine for Subclinical Hypothyroidism vs Placebo for Levothyroxine - Subclinical Hypothyroidism; Apgar at 1 min < 4; Test type: Superiority or Other; p = 0.76, Chi-squared
Statistical Analysis 2: Comparison: Levothyroxine for Hypothyroxinemia vs Placebo for Levothyroxine - Hypothyroxinemia; Apgar > 4 at 1 minute; Test type: Superiority or Other; p = 0.76, Chi-squared
Statistical Analysis 3: Comparison: Levothyroxine for Subclinical Hypothyroidism vs Placebo for Levothyroxine - Subclinical Hypothyroidism; Apgar < 7 at 5 minutes; Test type: Superiority or Other; p = 0.69, Chi-squared
Statistical Analysis 4: Comparison: Levothyroxine for Hypothyroxinemia vs Placebo for Levothyroxine - Hypothyroxinemia; Apgar < 7 at 5 minutes; Test type: Superiority or Other; p = 0.45, Chi-squared

18. Secondary Outcome: Number of Infants Admitted to NICU
Description: Admission to NICU
Time Frame: Delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Levothyroxine for Subclinical Hypothyroidism | Placebo for Levothyroxine - Subclinical Hypothyroidism | Levothyroxine for Hypothyroxinemia | Placebo for Levothyroxine - Hypothyroxinemia
Number analyzed (Participants) | 339 | 338 | 263 | 261
Participants | 29 | 21 | 31 | 31
Statistical Analysis 1: Comparison: Levothyroxine for Subclinical Hypothyroidism vs Placebo for Levothyroxine - Subclinical Hypothyroidism; Test type: Superiority or Other; p = 0.24, Chi-squared
Statistical Analysis 2: Comparison: Levothyroxine for Hypothyroxinemia vs Placebo for Levothyroxine - Hypothyroxinemia; Test type: Superiority or Other; p = 0.97, Chi-squared

19. Secondary Outcome: Infants With Birth Weight < 10th Percentile (Gestational Age z Score)
Description: Birth weight < 10th percentile (gestational age z score)
Time Frame: Delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Levothyroxine for Subclinical Hypothyroidism | Placebo for Levothyroxine - Subclinical Hypothyroidism | Levothyroxine for Hypothyroxinemia | Placebo for Levothyroxine - Hypothyroxinemia
Number analyzed (Participants) | 339 | 338 | 263 | 261
Participants | 33 | 27 | 23 | 20
Statistical Analysis 1: Comparison: Levothyroxine for Subclinical Hypothyroidism vs Placebo for Levothyroxine - Subclinical Hypothyroidism; Test type: Superiority or Other; p = 0.45, Chi-squared
Statistical Analysis 2: Comparison: Levothyroxine for Hypothyroxinemia vs Placebo for Levothyroxine - Hypothyroxinemia; Test type: Superiority or Other; p = 0.68, Chi-squared

20. Secondary Outcome: Neonatal Head Circumference (Centimeters)
Description: Neonatal head circumference measured within 24 hours of birth. This measurement is included based on a report showing that maternal treatment with thyroxine for overt hypothyroidism was associated with reduced head circumference in the newborn infant
Time Frame: Within 24 hours of birth
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Levothyroxine for Subclinical Hypothyroidism | Placebo for Levothyroxine - Subclinical Hypothyroidism | Levothyroxine for Hypothyroxinemia | Placebo for Levothyroxine - Hypothyroxinemia
Number analyzed (Participants) | 339 | 338 | 263 | 261
centimeters | 33.9 (1.8) | 33.9 (1.7) | 33.9 (1.8) | 34.2 (1.6)
Statistical Analysis 1: Comparison: Levothyroxine for Subclinical Hypothyroidism vs Placebo for Levothyroxine - Subclinical Hypothyroidism; Test type: Superiority or Other; p = 0.46, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Levothyroxine for Hypothyroxinemia vs Placebo for Levothyroxine - Hypothyroxinemia; Test type: Superiority or Other; p = 0.19, Wilcoxon (Mann-Whitney)

21. Secondary Outcome: Number of Infants With Respiratory Distress Syndrome
Description: Respiratory distress syndrome (RDS) will be defined based on a clinical diagnosis of RDS Type I and oxygen therapy (FiO2 ≥ 0.40) for greater than or equal to 24 hours. For infants dying before 24 hours of age, a clinical diagnosis of RDS Type I and oxygen therapy (FiO2 ≥ 0.40) are sufficient.
Time Frame: Delivery and greater than or equal to 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Levothyroxine for Subclinical Hypothyroidism | Placebo for Levothyroxine - Subclinical Hypothyroidism | Levothyroxine for Hypothyroxinemia | Placebo for Levothyroxine - Hypothyroxinemia
Number analyzed (Participants) | 339 | 338 | 263 | 261
Participants | 9 | 6 | 4 | 5
Statistical Analysis 1: Comparison: Levothyroxine for Subclinical Hypothyroidism vs Placebo for Levothyroxine - Subclinical Hypothyroidism; Test type: Superiority or Other; p = 0.45, Chi-squared
Statistical Analysis 2: Comparison: Levothyroxine for Hypothyroxinemia vs Placebo for Levothyroxine - Hypothyroxinemia; Test type: Superiority or Other; p = 0.75, Chi-squared

22. Secondary Outcome: Number of Infants With Retinopathy or Prematurity
Description: This diagnosis will be reached when an ophthalmologic examination of the retina has been performed and ROP is diagnosed at Stage I (demarcation line in the retina) or greater
Time Frame: Through 72 hours of birth
Measure: Count of Participants; unit: Participants
Arm/Group | Levothyroxine for Subclinical Hypothyroidism | Placebo for Levothyroxine - Subclinical Hypothyroidism | Levothyroxine for Hypothyroxinemia | Placebo for Levothyroxine - Hypothyroxinemia
Number analyzed (Participants) | 339 | 338 | 263 | 261
Participants | 1 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Levothyroxine for Subclinical Hypothyroidism vs Placebo for Levothyroxine - Subclinical Hypothyroidism; Test type: Superiority or Other; p = 1.00, Fisher Exact

23. Secondary Outcome: Number of Infants With Necrotizing Enterocolitis
Description: Necrotizing enterocolitis (NEC) is defined by the following: the unequivocal presence of intramural air on abdominal x-ray, perforation seen on abdominal x-ray, clinical evidence as suggested by erythema and induration of the abdominal wall, or intra-abdominal abscess formation, or stricture formation observed at surgery or autopsy following an episode of suspected NEC. The condition is classified based on the Bell staging system
Time Frame: Delivery within 2 weeks of birth
Measure: Count of Participants; unit: Participants
Arm/Group | Levothyroxine for Subclinical Hypothyroidism | Placebo for Levothyroxine - Subclinical Hypothyroidism | Levothyroxine for Hypothyroxinemia | Placebo for Levothyroxine - Hypothyroxinemia
Number analyzed (Participants) | 339 | 338 | 263 | 261
Participants | 1 | 1 | 2 | 0
Statistical Analysis 1: Comparison: Levothyroxine for Subclinical Hypothyroidism vs Placebo for Levothyroxine - Subclinical Hypothyroidism; Test type: Superiority or Other; p = 1.00, Fisher Exact
Statistical Analysis 2: Comparison: Levothyroxine for Hypothyroxinemia vs Placebo for Levothyroxine - Hypothyroxinemia; Test type: Superiority or Other; p = 0.50, Fisher Exact

24. Secondary Outcome: Number of Infants With Bronchopulmonary Dysplasia
Description: Bronchopulmonary dysplasia (BPD) is defined as the need for supplemental oxygen at 36 weeks corrected age, for babies born <34 weeks by project gestational age only
Time Frame: Through 72 hours post delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Levothyroxine for Subclinical Hypothyroidism | Placebo for Levothyroxine - Subclinical Hypothyroidism | Levothyroxine for Hypothyroxinemia | Placebo for Levothyroxine - Hypothyroxinemia
Number analyzed (Participants) | 339 | 338 | 263 | 261
Participants | 0 | 1 | 0 | 1
Statistical Analysis 1: Comparison: Levothyroxine for Subclinical Hypothyroidism vs Placebo for Levothyroxine - Subclinical Hypothyroidism; Test type: Superiority or Other; p = 0.50, Fisher Exact
Statistical Analysis 2: Comparison: Levothyroxine for Hypothyroxinemia vs Placebo for Levothyroxine - Hypothyroxinemia; Test type: Superiority or Other; p = 0.49, Fisher Exact

25. Secondary Outcome: Number of Infants With Respiratory Therapy Greater Than or Equal to 1 Day
Description: oxygen therapy (FiO2 ≥ 0.40) for greater than or equal to 24 hours
Time Frame: 72 hours post delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Levothyroxine for Subclinical Hypothyroidism | Placebo for Levothyroxine - Subclinical Hypothyroidism | Levothyroxine for Hypothyroxinemia | Placebo for Levothyroxine - Hypothyroxinemia
Number analyzed (Participants) | 339 | 338 | 263 | 261
Participants | 11 | 11 | 13 | 12
Statistical Analysis 1: Comparison: Levothyroxine for Subclinical Hypothyroidism vs Placebo for Levothyroxine - Subclinical Hypothyroidism; Test type: Superiority or Other; p = 0.99, Chi-squared
Statistical Analysis 2: Comparison: Levothyroxine for Hypothyroxinemia vs Placebo for Levothyroxine - Hypothyroxinemia; Test type: Superiority or Other; p = 0.85, Chi-squared

26. Secondary Outcome: Number of Days in the Hospital Nursery
Description: Median number of days in the hospital nursery
Time Frame: Through hospital discharge
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Levothyroxine for Subclinical Hypothyroidism | Placebo for Levothyroxine - Subclinical Hypothyroidism | Levothyroxine for Hypothyroxinemia | Placebo for Levothyroxine - Hypothyroxinemia
Number analyzed (Participants) | 339 | 338 | 263 | 261
days | 2 [2 to 2] | 2 [2 to 2] | 2 [2 to 2] | 2 [2 to 2]
Statistical Analysis 1: Comparison: Levothyroxine for Subclinical Hypothyroidism vs Placebo for Levothyroxine - Subclinical Hypothyroidism; Test type: Superiority or Other; p = 0.43, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Levothyroxine for Hypothyroxinemia vs Placebo for Levothyroxine - Hypothyroxinemia; Test type: Superiority or Other; p = 0.39, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Data on adverse events was collected for each participant beginning with enrollment through the final 5-year follow-up with the mother and child.
Description: The at-risk population for non-serious adverse events (side effects) was based on patients who had been seen for a least one study visit where side effect information was assessed, so the at-risk population for side effects varies from the total number of patients randomized and assessed for serious adverse events.
Groups:
- Placebo for Levothyroxine - Subclinincal Hypothyroidism: Placebo for Levothyroxine for participants with subclinical hypothyroidism
  Placebo for Levothyroxine
- Placebo for Levothyroxine: Placebo for Levothyroxine for participants with hypothyroxinemia
  Placebo for Levothyroxine
Arm/Group | Levothyroxine for Subclinical Hypothyroidism | Placebo for Levothyroxine - Subclinincal Hypothyroidism | Levothyroxine for Hypothyroxinemia - Hypothyroxinemia | Placebo for Levothyroxine
Serious Adverse Events (participants affected / at risk) | 4/339 | 2/338 | 3/265 | 2/261
Other Adverse Events (participants affected / at risk) | 51/338 | 41/336 | 25/261 | 34/259
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levothyroxine for Subclinical Hypothyroidism (N=339) | Placebo for Levothyroxine - Subclinincal Hypothyroidism (N=338) | Levothyroxine for Hypothyroxinemia - Hypothyroxinemia (N=265) | Placebo for Levothyroxine (N=261)
Maternal atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hashimoto's thryoiditis (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest/abdominal pain (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Maternal death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Maternal death at 2 years postpartum
Irregular fetal heart rate (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
IUGR, non-reassuring (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Non-reassuring Intrauterine Growth Restriction
Abnormal Doppler (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neonatal Hypoxic-Ischemic Encephalopathy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Hypoxic-Ischemic Encephalopathy
Autism Spectrum Disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neonatal Severe Hearing Loss (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Levothyroxine for Subclinical Hypothyroidism (N=338) | Placebo for Levothyroxine - Subclinincal Hypothyroidism (N=336) | Levothyroxine for Hypothyroxinemia - Hypothyroxinemia (N=261) | Placebo for Levothyroxine (N=259)
Vomiting/Nausea (Gastrointestinal disorders) | 18 | 8 | 10 | 15 — Participant reported side effect
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 2 | 2 — Participant reported side effect
Nervousness (General disorders) | 4 | 3 | 2 | 2 — Participant reported side effect
Fatigue (General disorders) | 4 | 4 | 4 | 5 — Participant reported side effect
Headaches (General disorders) | 10 | 8 | 3 | 4 — Participant reported side effect
Other side effects (General disorders) | 18 | 13 | 4 | 10 — Participant reported side effects including allergic reaction.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes